CLINICAL TRIAL: NCT02024100
Title: Observational Study to Investigate the Effectiveness of Eprosartan on Pulse Pressure in Hypertensive Patients With Metabolic Syndrome
Brief Title: Observational Study to Investigate the Effectiveness of Eprosartan on Pulse Pressure (Teveten_MS)
Status: Completed | Type: Observational
Sponsor: Handok Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HD_EPR_OS2013
Record Dates: First submitted 2013-12-26; First posted 2013-12-31 (Estimated); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study is to identify the effectiveness of Eprosartan on pulse pressure in hypertensive patients with metabolic syndrome

-Definition of pulse pressure (PP): Difference between systolic and diastolic blood pressure produced one heart beat.

DETAILED DESCRIPTION:
Primary Objective

-To assess the changes of pulse pressure at 12 weeks

Secondary Objectives

* To assess the changes of pulse pressure at 4, 24 weeks
* To assess the changes of systolic blood pressure and diastolic blood pressure at each visit
* Percentage of responder rate* at each visit and time to get normalized BP from enrollment
* Responder rate at last visit
* To assess IIEF-5 (5-item Version of the International Index of Erectile Function) score at enrollment and 24 weeks (percentage of patients with ED according to IIEF-5, Changes of IIEF-5 domains)
* Percentage of patients with erectile dysfunction (ED) according to IIEF-5 and changes of PP in subgroup (age 65, body mass index (BMI) 23, diabetes mellitus, dyslipidemia, benign prostate hypertrophy)
* Analysis of correlation between ED and concomitant disease and concomitant medications in patients who received Eprosartan
* Score changes of Framingham 10-year Coronary Heart Disease (CHD) risk at 1st visit, 4th visit
* Percentages of Eprosartan monotherapy and multiple antihypertensive therapies at enrollment and last visit
* Reason for treatment discontinuation (Inadequate BP control, adverse events, others)
* Adverse events

  * Responder rate: SBP <140mmHg and DBP <90mmHg (SBP <140mmHg and DBP <85mmHg for patients with diabetes mellitus)

ELIGIBILITY:
Inclusion Criteria:

1. 20-80 years old patient at the 1st visit
2. Patient who is determined to prescribe Eprosartan for hypertension (patient with at least one of the following conditions) (1) Newly diagnosed hypertension (2) Inability to tolerate hypertension (for example: adverse event) (3) Lack of response to current antihypertensive medications
3. Metabolic syndrome patient (fulfill 3 or more components before enrollment) (1) Waist circumference (>90 for men, >80 for women) (2) Triglycerides (≥150mg/dl) (3) HDL cholesterol (<40mg/dl for men, <50mg/dl for women) (4) SBP≥130mmHg or DBP≥85mmHg or on antihypertensive medications) (5) Fasting glucose level (≥100mg/dl) or on antidiabetic medications

   * MS diagnosis origin: Korean diabetes association

Exclusion Criteria:

1. Patients who is administered with 3 or more than 3 antihypertensive drugs
2. Patients who is contraindicated with Eprosartan by the product label

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General hospitals
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2014-02-06 (Actual); Primary Completion 2016-12-26 (Actual); Study Completion 2016-12-26 (Actual)

PRIMARY OUTCOMES:
To assess the changes of pulse pressure at 12 weeks | 12 weeks
  Calculating pulse pressure at 3rd(12weeks) visit and it will be presented in descriptive statistics quantity

SECONDARY OUTCOMES:
- changes of pulse pressure at 4, 24 weeks - changes of blood pressure at 4, 12, 24 weeks - Duration to get normalized BP - assess IIEF-5 score - Score changes of Framingham 10-year CHD risk | 24 weeks
  * Calculating pulse pressure at each visit and it will be presented in descriptive statistics quantity
  * Variation of the pulse pressure at each visit will be presented in descriptive statistics quantity and average variation's 95% confidence interval will be calculated
  * Calculating systolic blood pressure and diastolic blood pressure at each visit and it will be presented in descriptive statistics quantity
  * Severity of erectile dysfunction will be presented a contingency table and symmetry testing will be done whether there is a significant difference in the data
  * As sub-analysis, type of study drug, age, BMI, with/without diabetes mellitus, with/without dyslipidemia, with/without benign prostate hypertrophy, type of treatment will be considered
  * For safety analysis, overall incidence rate of adverse event will be presented and frequency and percentage will be presented according to body organs and preferable terminology

CONTACTS AND LOCATIONS:
Overall Officials: Chang Hwan Yoon, MD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Bundang-gu, South Korea